CLINICAL TRIAL: NCT03293680
Title: Survival, Quality of Life and Self-reported Outcomes of Elderly Patients With Advanced Non-small Cell Lung Cancer Treated With Pembrolizumab (MK-3475) in the First Line Setting
Brief Title: Pembrolizumab in Elderly Patients With Advanced Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GECP 16/06_PEBEL
Record Dates: First submitted 2017-09-19; First posted 2017-09-26 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab Arm (Experimental): 1 group, Pembrolizumab (MK-3475) 200 mg, every 3 weeks
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab (MK-3475) 200 mg, every 3 weeks
  Other Names: KEYTRUDA

SUMMARY:
This is a multi-center phase II trial of intravenous (IV) Pembrolizumab MK-3475 in subjects older than 70 years with advanced Non-small cell Lung Cancer (NSCLC) expressing Programmed death-ligand 1 (PD-L1). 82 patients will be enrolled in this trial to examine the efficacy, the impact on geriatric assessments, the quality of life and the self-reported outcomes.

DETAILED DESCRIPTION:
Subjects will receive MK-3475 at a fixed dose of 200 mg every 3 weeks (Q3W) (Figure 1). Subjects will be evaluated every 9 weeks (63 ± 7 days) with radiographic imaging to assess response to treatment. QoL and Self-reported Health Questionnaires, as well as geriatric follow-up will be performed at the same intervals. Investigators will make all treatment-based decisions using immune-related Response Criteria (irRC). However, for determination of overall response rate (ORR) and progression-free survival (PFS), the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 will be used. Adverse events will be monitored throughout the trial and graded in severity according to the guidelines outlined in the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Treatment with MK-3475 will continue until two years of therapy have been administered, documented disease progression, unacceptable adverse event(s), intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, subject withdraws consent, noncompliance with trial treatment or procedure requirements, or administrative reasons.

After the end of treatment, each subject will be followed for a minimum of 30 days for adverse event monitoring (serious adverse events will be collected for up to 90 days after the end of treatment unless the subject starts a new anticancer therapy between days 31 and 90). Subjects will have post-treatment follow-up for disease status, including initiating a non-study cancer treatment and experiencing disease progression, until death, withdrawing consent, or becoming lost to follow-up.

Participation in this trial will be dependent upon supplying tumor tissue from a newly obtained formalin-fixed specimen from locations not radiated prior to biopsy. The specimen will be evaluated at a central laboratory facility for expression status of Programmed death-ligand 1(PD-L1) in a prospective manner. Only subjects whose tumors express Programmed death-ligand 1(PD-L1) as determined by the central laboratory facility will be eligible for inclusion in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histological or cytological documented stage III B or IV squamous and non-squamous non-small-cell lung cancer previously untreated.
2. Epidermal Growth Factor receptor (EGFR) and Anaplastic lymphoma kinase (ALK) have to be wild-type.
3. The subject must be willing and able to provide written informed consent/assent for the trial.
4. Patients must be aged more than 70 years, on day of signing informed consent.
5. Measurable disease (at least 1 lesion) based on RECIST criteria v1.1. Patients will not be eligible if this lesion was irradiated before inclusion.
6. Be willing to provide tissue from a newly obtained core or excision biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
7. PD-L1 expression ≥ 1%
8. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group Performance Scale.
9. Screening laboratory values must meet the following criteria (Table 1, see protocol), all screening laboratory tests should be performed within 8 days of treatment initiation.
10. Male subjects of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy at a dose over 10 mg of prednisone or equivalent, or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active Tuberculosis Bacillus
4. Hypersensitivity to Pembrolizumab or any of its excipients.
5. Has had any prior anti-cancer therapy for his or her metastatic NSCLC. In the case of patients who have progressed to a metastatic stage after having been treated for early stage NSCLC, chemotherapy or radiation therapy as part of this previous treatment is allowed, provided they have been completed more than three months ago. Patients who received adjuvant or neoadjuvant treatment or both for early stages will be eligible for this trial. All adverse events related to these previous treatments must have recovered (i.e., ≤ Grade 1 or at baseline).
6. Has had any previous malignancy (except non melanoma skin cancer, and cancer in situ of: bladder, gastric, colon, cervical/dysplasia, melanoma, breast), unless a complete remission was achieved at least 2 years prior to study entry and no additional therapy is required or anticipated to be required during the study period.
7. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate if they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids at a dose over 10 mg of prednisone or equivalent, for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
8. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxin, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
9. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
10. Has an active infection requiring systemic therapy.
11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
13. Has any geriatric exclusion criteria:

    * advanced dementia (GDS ranking >6)
    * moderate or severe functional dependence (Barthel Index < 35)
    * Life expectancy less than one year, due to co-morbidities other than lung cancer.
14. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
15. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., Hepatitis C Virus RNA [qualitative] is detected).
16. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
17. Evidence of interstitial lung disease.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Remei Blanco, PhD, Principal Investigator — Hospital de Terrassa
Locations (12):
- Spain (12):
  - ICO-Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital Universitario Sta Lucia, Cartagena, Murcia
  - Hospital Lluís Alcanyís, Xàtiva, Valencia
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Virgen de la Luz, Cuenca
  - Hospital Lucus Agustí, Lugo
  - Fundación Jiménez Díaz, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Dr. Peset, Valencia
  - Hospital La Fe, Valencia
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org
- See also: Lung Cancer Publication — https://doi.org/10.1016/j.lungcan.2023.107318

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 83 patients were recruited between January 2017 and November 2019 and 82 patients received treatment. Of these, 74 patients were finally analysed since eight were inclusion errors.
Period: Overall Study
Arm/Group | Pembrolizumab Arm
Started | 83
Completed | 74
Not Completed | 9
Not completed — Death | 1
Not completed — Did not meet inclusion criteria | 8

BASELINE CHARACTERISTICS:
Population: We performed the analyses on the intention-to-treat (ITT) population.
Arm/Group | Pembrolizumab Arm
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.1 (5.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 74
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Spain | 74
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 32
  Squamous | 33
  Large cell carcinoma | 2
  Aden squamous | 1
  Not otherwise specified / Undifferentiated | 6
Current cancer stage [Count of Participants; unit: Participants] — Staging is a classification where cancer is located, if or where it has spread and whether it's affecting other parts of the body.
  There are 5 stages for NSCLC:
  Stage 0:tumor hasn't grown into nearby normal lung tissues Stage I:small tumor that hasn't spread to any lymph nodes Stage II: medium tumor that hasn't spread to the nearby lymph nodes or N1 Stage III: cancer spread to the lymph nodes but haven't spread to other distant parts of the body Stage IV:cancer has spread to more than 1 area in the other lung, the fluid surrounding the lung or the heart, or distant parts of the body
  Participants
    IIIB | 6
    IV | 68
Previous antineoplastic treatments [Number; unit: participants]
  Radiotherapy | 24
  Surgery | 9
  Adjuvant chemotherapy | 6
  Concurrent chemoradiotherapy | 5
  Neo-adjuvant chemotherapy | 2
  No therapy | 28
PD-L1 [Count of Participants; unit: Participants] — Only subjects whose tumors demonstrate evidence of PD-L1 expression (on the neoplastic cells) are eligible for enrollment. Positivity is defined as at least 1% of tumour cells expressing PD-L1 on histochemistry (i.e., a tumour proportion score ≥1%).
  Participants
    1-19% | 16
    20-49% | 23
    ≥50% | 35
ECOG performance Status at diagnosis [Count of Participants; unit: Participants] — ECOG Performance Status Scale: It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability
  GRADES:
  ECOG 0: Fully active. ECOG 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature ECOG 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours ECOG 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours ECOG 4: Completely disabled
  Participants
    ECOG 0 | 18
    ECOG 1 | 56
Smoking history [Count of Participants; unit: Participants]
  Never (≤100 cigarettes/lifetime) | 11
  Former smoker (≥1 year) | 51
  Current smoker | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Defined as the length of time from either the date of diagnosis or the start of the treatment that patients diagnosed with the disease are still alive.
Time Frame: From the date of inclusion of the first patient to until end of follow up, up to 36 months.
Population: We performed the analyses on the intention-to-treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Arm
Number analyzed (Participants) | 74
Months | 19.2 [11.3 to 25.5]

2. Secondary Outcome: Changes in Health-related Quality of Life With Lung Cancer Symptom Scale
Description: To evaluate changes in health-related quality of life in responder and non-responder patients older than 70 years with advanced non-small cell lung cancer. QLQ-C30 Quality of Life Questionnaire. The EORTC Core Quality of Life questionnaire (EORTC QLQ-C30) is designed to measure cancer patients' physical, psychological and social functions. The questionnaire is composed of multi-item scales and single items.
  All EORTC QLQ-C30 scale scores range from 0 to 100. A high score for a functional scale represents a high level of functioning, whereas a high score for a symptom scale/single item represents a high level of symptom- atology
Time Frame: Beginning of cycle 1 (week 1) and beginning of cycle 18 (week 54) (each cycle is 3 weeks)
Population: Intention to treat population
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Pembrolizumab Arm
Number analyzed (Participants) | 74
units on a scale
  At the beginning of the first cycle | 66.7 [16.7 to 100]
  At the beginning of the eighteenth cycle | 92.3 [72.3 to 100]

3. Secondary Outcome: Impact on Functional Assessments Measured With Barthel Scale
Description: To evaluate the impact on functional geriatric assessments of patients older than 70 years with advanced non-small cell lung cancer. The Barthel Index assesses activities in two major categories: Personal care and mobility. The personal care items include tasks such as drinking from a cup, dressing, grooming, bathing, and bowel and bladder continence. The scoring is as follows: scores of 0-20 indicate "total" dependency. scores of 21-60 indicate "severe" dependency. scores of 61-90 indicate "moderate" dependency. scores of 91-99 indicate "slight" dependency, score of 100 indicate independent.
Time Frame: Beginning of cycle 1 (week 1), beginning of cycle 4 (week 12), beginning of cycle 7 (week 21), beginning of cycle 10 (week 30), beginning of cycle 13 (week 39), beginning of cycle 16 (week 48) and beginning of cycle 18 (week 54) (each cycle is 3 weeks)
Population: Intention to treat population
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Pembrolizumab Arm
Number analyzed (Participants) | 74
units on a scale
  At the beginning of Cycle 1 | 100 [50 to 100]
  At the beginning of Cycle 4 | 100 [76 to 100]
  At the beginning of Cycle 7 | 100 [65 to 100]
  At the beginning of Cycle 10 | 100 [75 to 100]
  At the beginning of Cycle 13 | 100 [70 to 100]
  At the beginning of Cycle 16 | 100 [58 to 100]
  At the beginning of Cycle 18 | 97 [90 to 100]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: To describe Progression-free Survival (PFS), according to RECIST criteria v. 1.1 of the first-line treatment with pembrolizumab (MK-3475) in elderly patients with advanced NSCLC. PFS defined as the length of time from the date of randomization to the date of the first documented progression of disease. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From the inclusion date in the study until first progression or end of follow up, up to 36 months
Population: It is performed the analyses on the intention-to-treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Arm
Number analyzed (Participants) | 74
Months | 6.1 [4.6 to 8.6]

5. Secondary Outcome: Overall Survival Rate at 2 Years.
Description: To evaluate the overall survival percentage of the patients included at two years
Time Frame: From the date of inclusion of the first patient until two years follow up visit, up to 24 months
Population: Intention to treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab Arm
Number analyzed (Participants) | 74
percentage of participants | 40.2 [28.6 to 51.5]

6. Secondary Outcome: OS for Patients With a PD-L1 Under 50%
Description: Defined as the length of time from the date of the start of the treatment that patients diagnosed with the disease and PD¨-L1 under 50% are still alive.
Time Frame: From the initiation of treatment until end of follow up, up to 36 months
Population: It is performed the analyses on the intention-to-treat (ITT) population.
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Arm
Number analyzed (Participants) | 39
Months | 16.5 [6.8 to 24.6]

7. Secondary Outcome: OS for Patients With a PD-L1 Greater Than or Equal to 50%
Description: Defined as the length of time from the start of the treatment that patients diagnosed with the disease and PD-L1 greater than or equal to 50% are still alive.
Time Frame: From the initiation of treatment until end of follow up, up to 36 months
Population: It is performed the analyses on the intention-to-treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Arm
Number analyzed (Participants) | 35
Months | 23.3 [14.8 to 36]

ADVERSE EVENTS:
Time Frame: 36 months
Description: The severity of AE will be determined using CTCAE version 4.03
Arm/Group | Pembrolizumab Arm
All-Cause Mortality (participants affected / at risk) | 46/74
Serious Adverse Events (participants affected / at risk) | 46/74
Other Adverse Events (participants affected / at risk) | 59/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab Arm (N=74)
Progression disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 36 (36)
Other causes of death (General disorders) | 10 (10)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab Arm (N=74)
Platelet count decreased (Investigations) | 6 (6)
Increased creatinine level (Investigations) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Fatigue (General disorders) | 23 (23)
Diarrhoea (Gastrointestinal disorders) | 14 (14)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 19 (19)
Rash (Skin and subcutaneous tissue disorders) | 11 (11)
Hyperthyroidism (Endocrine disorders) | 9 (9)
Hypothyroidism (Skin and subcutaneous tissue disorders) | 7 (7)
Anorexia (Metabolism and nutrition disorders) | 12 (12)

LIMITATIONS AND CAVEATS:
Age-specific issues for complete the study relative to older cancer patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT03293680/Prot_SAP_000.pdf